CLINICAL TRIAL: NCT06193252
Title: Slow-SPEED-NL: Slowing Parkinson's Early Through Exercise Dosage-Netherlands
Acronym: Slow-SPEED-NL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Stichting ParkinsonNL (Unknown); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Michael J. Fox Foundation for Parkinson's Research (Other); Parkinson's UK (Other); Cure Parkinson's (Other); Edmond J. Safra Foundation (Unknown); Davis Phinney Foundation (Other); Donders Centre for Cognitive Neuroimaging (Other); Anne Wojcicki Foundation (Unknown); Sleep Medicine Centre Kempenhaeghe (Other); Sleep Medicine Centre SEIN (Unknown); Queen Mary University of London (Other); 23andMe, Inc. (Industry); Parkinsons Progression Markers Initiative (PPMI) (Unknown); Massachusetts General Hospital (Other); Harvard School of Public Health (HSPH) (Other); IJsfontein B.V., Netherlands (Unknown); Hoffmann-La Roche (Industry); Erasmus Medical Center (Other); University of Illinois at Chicago (Other); University of Rochester (Other); University of Bristol (Other); University of Plymouth (Other); University of Luebeck (Other); McGill University (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NL84072.091.23
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease; Prodromal Stage; Neurodegenerative Diseases; Parkinsonian Disorders; REM Sleep Behavior Disorder; Basal Ganglia Diseases; Central Nervous System Diseases; Synucleinopathies; Nervous System Diseases; Cerebral Disorder; Brain Diseases
Keywords: Physical Activity; Prevention; Remote; Mobile Health (mHealth); Feasibility; Exercise; Digital biomarker; Blood; Imaging; MRI; Motivational application; Walking; Parkinson Disease; Prodromal
MeSH Terms: conditions — Parkinson Disease; Prodromal Symptoms; Neurodegenerative Diseases; Parkinsonian Disorders; REM Sleep Behavior Disorder; Basal Ganglia Diseases; Central Nervous System Diseases; Synucleinopathies; Nervous System Diseases; Brain Diseases; Motor Activity

STUDY DESIGN:
Intervention Model Description: Double-blind randomized controlled trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Large proportional increase in step count and minutes exerting moderate to vigorous physical activity (MVPA) relative to baseline level.
  Interventions: Behavioral: Increase of physical activity volume and intensity with the use of a motivational smartphone application
- Active control (Active Comparator): Small proportional increase in step count and minute exerting moderate to vigorous physical activity (MVPA) relative to baseline level.
  Interventions: Behavioral: Increase of physical activity volume and intensity with the use of a motivational smartphone application

INTERVENTIONS:
Behavioral: Increase of physical activity volume and intensity with the use of a motivational smartphone application — A motivational smartphone application will be available for all participants using their own smartphone: the Slow-SPEED app. The Slow-SPEED app will motivate participants to increase the volume and intensity of their physical activity in daily life over a long period of time (2 years) based on their own baseline levels. Different treatment arms will receive different physical activity goals. The app offers participants feedback and support, that will stimulate them to reach their individual physical activity goal (i.e. incremental relative increase of step count and minutes exerting ≥ 64% of maximum heart rate reflecting MVPA relative to baseline level.).

SUMMARY:
The goal of this clinical trial is to investigate the feasibility if a remotely administered smartphone app can increase the volume and intensity of physical activity in daily life in patients with isolated Rapid Eye Movement (REM) sleep behaviour disorder over a long period of time (24 months).

Participants will be tasked to achieve an incremental increase of daily steps (volume) and amount of minutes exercised at a certain heart rate (intensity) with respect to their own baseline level. Motivation with regards to physical activity will entirely be communicated through the study specific Slow Speed smartphone app. Primary outcomes will be compliance expressed as longitudinal change in digital measures of physical activity (step count) measured using a Fitbit smartwatch. Exploratory outcomes entail retention rate, completeness of remote digital biomarker assessments, digital prodromal motor and non-motor features of PD, blood biomarkers and brain imaging markers. Using these biomarkers, we aim to develop a composite score (prodromal load score) to estimate the total prodromal load. An international exercise study with fellow researchers in the United States and United Kingdom are currently in preparation (Slow-SPEED). Our intention is to analyse overlapping outcomes combined where possible through a meta-analysis plan, to obtain insight on (determinants of) heterogeneity in compliance and possible efficacy across subgroups

DETAILED DESCRIPTION:
Rationale: Parkinson's Disease (PD) is the fastest growing neurodegenerative disease. Exercise beneficially effects motor symptoms and neuroplasticity in people with PD. However, disease-slowing interventions have been ineffective in clinically manifest PD, when pathology is already advanced, but could succeed in prodromal PD, when pathology is limited. People with an isolated Rapid Eye Movement (REM) sleep Behaviour Disorder (iRBD) have a high risk to develop clinically manifest PD or a related neurodegenerative disease and are therefore considered to have probable prodromal PD. This study will take an important step forward by studying the feasibility and preliminary efficacy of long-term physical activity on prodromal symptoms and disease progression in people with probable prodromal PD using a newly developed, fully remote smartphone-based app. The app is inspired by the app used in the STEPWISE trial (NCT04848077).

Objective: The goal of this clinical trial is to investigate whether a smartphone app can increase the volume and intensity of physical activity in daily life in patients with iRBD at risk of developing PD for a long period of time (24 months). The secondary aim is the potential group effect on physical fitness, digital prodromal motor- and non-motor symptoms. Thirdly, we investigate whether the intervention, prodromal motor- and non-motor symptoms can be assessed remotely in a digital, decentralized fashion. Fourthly, we aim to investigate the effect on imaging- and fluid biomarkers to identify markers for prodromal progression. Using these biomarkers, we aim to develop a composite score (prodromal load score) to estimate the total prodromal load.

The anticipated fluid biomarkers outcomes are subject to potential alterations in the event of the development and implementation of novel techniques and/or biomarkers during the course of this study.

Study design: Double-blind randomized controlled trial

Study population: A total of 110 Dutch patients with iRBD (ICSD-3 criteria) aged 50 years and older, who are in possession of a suitable smartphone without mobility hampering conditions and absence of cognitive impairment which impedes usage of a smartphone will be recruited

Intervention: Participants will be randomized to a group and will be motivated to increase the volume and intensity of physical activity based on their own baseline level. The groups differ in the amount of physical activity that they are tasked to achieve.

ELIGIBILITY:
Inclusion Criteria:

* previously diagnosed with iRBD meeting the following criteria according to the International Classification of Sleep Disorders (ICSD-3)
* able to understand the Dutch language
* being able to walk independently inside the home without the use of a walking aid
* Not in a high physical activity range during the 4-week eligibility and baseline period
* in possession of a suitable smartphone compatible with the Slow-SPEED app, the Fitbit app and the Roche PD Research Mobile application.

Exclusion Criteria:

* clinically diagnosed or self-reported diagnosis neurodegenerative disease;
* self-reported weekly falls in the previous 3 months;
* dexterity problems or cognitive impairments hampering smartphone use;
* if they do not wish to be informed about an increased risk of developing diseases associated with iRBD
* if individual is not community-dwelling

Exclusion criteria for MRI only:

* history of epilepsy, structural brain abnormalities (i.e. stroke, traumatic defects, large arachnoid cysts) or brain surgery
* claustrophobia
* implanted electrical devices (i.e. pacemaker, deep-brain stimulator (DBS), neurostimulator)
* metal implants (such as prosthetics, ossicle prosthesis, metal plates or other non-removable metal part) or metal splinters
* pregnancy
* fear for incidental finding

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in step count per day | All 4 week periods between and including week -4 until 0 (baseline period) and week 100 until 104 (follow-up period)
  Mean change in step count per day as measured continuously with a smartwatch. Mean steps per day will be calculated from 4-week periods. Higher positive change in step count indicate more volume of physical activity.

SECONDARY OUTCOMES:
Change in moderate to vigorous physical activity (MVPA) per day | All 4 week periods between and including week -4 until 0 (baseline period) and week 100 until 104 (follow-up period)
  Change in number of minutes exerting (minimally) ≥ 64% of maximum heart rate, reflecting moderate intense physical activity, measured continuously using a smartwatch. Mean minutes per day will be calculated from 4-week periods. Higher positive change in minutes of MVPA indicate more aerobic physical activity.
Change in resting heart rate (physical fitness) | All 4 week periods between and including week -4 until 0 (baseline period) and week 100 until 104 (follow-up period)
  Change in resting heart rate per day as measured continuously with a smartwatch. Mean resting heart rate per day will be calculated from 4-week periods. Higher negative change (i.e. lower resting heart rate) indicate better function.
Change in heart rate variability (physical fitness) | All 4 week periods between and including week -4 until 0 (baseline period) and week 100 until 104 (follow-up period)
  Change in heart rate variability in Root Mean Square of Successive Differences (RMSSD) measured every 5 minutes with a smartwatch. Mean RMSSD per day will be calculated from 4-week periods. Higher positive change in RMSSD indicate better function.
Change in blood pressure (physical fitness) | Week 0 (baseline) and week 104 (follow-up)
  Change from baseline (week 0) blood pressure in mmHg assessed by a sphygmomanometer at follow-up (week 104). Lower scores indicate better function.
Change in VO2max (physical fitness) | All 4 week periods between and including week -4 until 0 (baseline period) and week 100 until 104 (follow-up period)
  Change in VO2max in ml/kg/min measured per day with a smartwatch. Mean VO2max per day will be calculated from 4-week periods. Higher positive change in VO2max indicate better function.
Change in heart rate variability (autonomic function) | All 4 week periods between and including week -4 until 0 (baseline period) and week 100 until 104 (follow-up period)
  Mean change in heart rate variability in Root Mean Square of Successive Differences (RMSSD) measured every 5 minutes with a smartwatch. Mean RMSSD per day will be calculated from 4-week periods. Higher positive change in RMSSD indicate better function.
Change in orthostatic blood pressure (autonomic function) | Week 0 (baseline) and week 104 (follow-up)
  Change in baseline (week 0) difference between supine and standing blood pressure measured with a sphygmomanometer to follow-up (week 104). Higher change indicate more autonomic dysfunction.
Change in anxiety and depression (HADS) | Week 0 (baseline), week 52 (1 year), week 104 (follow-up)
  Change from baseline (week 0) on the Hospital Anxiety and Depression Scale (HADS) at week 52 (1 year) and week 104 (follow-up). Range 0-42. Higher scores indicate worse function.
Change in cognition (MoCA) | Week 0 (baseline), week 104 (follow-up)
  Change from baseline (week 0) on the Montreal Cognitive Assessment (MoCA) at week 104 (follow-up). Range 0-30. Higher scores indicate better function.
Mean change in light sleep (sleep stage) | All 4 week periods between and including week -4 until 0 (baseline period) and week 100 until 104 (follow-up period)
  Mean change in light sleep stage measured continuously with a smartwatch. Mean duration of light sleep per day will be calculated from 4-week periods. Higher positive change indicate more light sleep.
Mean change in deep sleep (sleep stage) | All 4 week periods between and including week -4 until 0 (baseline period) and week 100 until 104 (follow-up period)
  Mean change in deep sleep stage measured continuously with a smartwatch. Mean duration of deep sleep per day will be calculated from 4-week periods. Higher positive change indicate more deep sleep.
Mean change in REM sleep (sleep stage) | All 4 week periods between and including week -4 until 0 (baseline period) and week 100 until 104 (follow-up period)
  Mean change in rapid eye movement (REM) sleep stage measured continuously with a smartwatch. Mean duration of REM sleep per day will be calculated from 4-week periods. Higher positive change indicate more REM sleep.
Change in self-reported sleep quality (PSQI) | Week 0 (baseline), week 52 (1 year), week 104 (follow-up)
  Change from baseline (week 0) on the Pittsburgh Sleep Quality Index (PSQI) at week 52 (1 year) and week 104 (follow-up). Range 0-21. Higher scores indicate worse sleep quality.
Change in olfaction (UPSIT) | Week 0 (baseline), week 104 (follow-up)
  Change from baseline (week 0) on the University of Pennsylvania Smell Identification Test (UPSIT) at week 104 (follow-up). Range 0-40. Higher scores indicate better function.
Change in motor symptoms (Roche PD Research mobile application) | Week 0 (baseline), week 6, week 12, week 18, week 24, week 30, week 36, week 42, week 48, week 54, week 60, week 66, week 72, week 78, week 84, week 90, week 96, week 102
  Change in motor symptoms measured digitally with the smartphone using the Roche PD Research mobile application. Higher scores indicate worse function.
Change in metabolism (blood based biomarkers) | Week 0 (baseline), week 26 (optional), week 52 (optional), week 78 (optional) and week 104 (follow-up)
  Change from baseline (week 0) on glucose and HbA1c at follow-up (week 104). Optional at week 26, week 52 and week 78. Lower scores indicate better metabolism.
Change in inflammation (blood based biomarkers) | Week 0 (baseline), week 26 (optional), week 52 (optional), week 78 (optional) and week 104 (follow-up)
  Change from baseline (week 0) on Tumor Necrosis Factor-α, Interleukin-6 (IL-6), IL-18, IGF-1, clusterin, Il-10, PGC-α (irisin) at follow-up (week 104). Optional at week 26, week 52 and week 78. Lower inflammatory markers indicate less inflammation. Higher anti-inflammatory markers indicate less inflammation.
Change in growth factors (blood based biomarkers) | Week 0 (baseline), week 26 (optional), week 52 (optional), week 78 (optional) and week 104 (follow-up)
  Change from baseline (week 0) on brain-derived neurotrophic factor (BDNF), Glial cell line-derived neurotrophic factor (GDNF), Platelet-derived growth factor (PDGF), Growth/differentiation factor 15 (GDF15) and Epidermal growth factor (EGF) at follow-up (week 104). Optional at week 26, week 52 and week 78. Higher growth factors indicate better function.
Change in ageing mechanism (blood based biomarkers) | Week 0 (baseline), week 26 (optional), week 52 (optional), week 78 (optional) and week 104 (follow-up)
  Change from baseline (week 0) on klotho at follow-up (week 104). Optional at week 26, week 52 and week 78. High ageing marker indicate better function (i.e. less aging)
Change in pathological protein (blood based biomarkers) | Week 0 (baseline), week 26 (optional), week 52 (optional), week 78 (optional) and week 104 (follow-up)
  Change from baseline (week 0) on α-synuclein at follow-up (week 104). Optional at week 26, week 52 and week 78. Low pathological protein indicate better function (i.e. less pathological process).
Change in neurodegeneration (blood based biomarkers) | Week 0 (baseline), week 26 (optional), week 52 (optional), week 78 (optional) and week 104 (follow-up)
  Change from baseline (week 0) on Neurofilament light (NfL) at follow-up (week 104). Optional at week 26, week 52 and week 78. Lower neurodegeneration markers indicate less neurodegeneration.
Change in brain volume (imaging biomarkers) | Week 0 (baseline) and week 104 (follow-up)
  Change from baseline (week 0) on T1 Voxel-Based-Morphometry (VBM) at follow-up (week 104). Higher scores indicate higher volume.
Change in white matter hyperintensities (imaging biomarkers) | Week 0 (baseline) and week 104 (follow-up)
  Change from baseline (week 0) on FLAIR at follow-up (week 104). Higher scores indicate worse status.
Change in basal ganglia; cortex [1] (imaging biomarkers) | Week 0 (baseline) and week 104 (follow-up)
  Change from baseline (week 0) on resting-state functional MRI (Rs-fMRI) at follow-up (week 104). Higher scores indicate better functional connectivity.
Change in basal ganglia; cortex [2] (imaging biomarkers) | Week 0 (baseline) and week 104 (follow-up)
  Change from baseline (week 0) on task-based functional MRI at follow-up (week 104). Higher scores indicate better functional connectivity.
Change in substantia nigra [1] (imaging biomarkers) | Week 0 (baseline) and week 104 (follow-up)
  Change from baseline (week 0) on diffusion tensor imaging (DTI) at follow-up (week 104). Higher scores indicate better tissue integrity.
Change in substantia nigra [2] (imaging biomarkers) | Week 0 (baseline) and week 104 (follow-up)
  Change from baseline (week 0) on Quantitative Susceptibility Mapping (QSM) at follow-up (week 104). Higher scores indicate more iron loading.
Change in substantia nigra [3]; locus coeruleus (imaging biomarkers) | Week 0 (baseline) and week 104 (follow-up)
  Change from baseline (week 0) on neuromelanin at follow-up (week 104). Higher scores indicate better tissue integrity.
Change in instrumental activities of daily living (ADL) (functional status) | Week 0 (baseline), week 52 (1 year) and week 104 (follow-up)
  Change from baseline (week 0) on Lawton instrumental ADL (iADL) scale at week 52 (1 year) and 104 (follow-up). Range 0-14. Higher score indicate better function.
Change in WHOQoL-BREF (quality of life) | Week 0 (baseline), week 52 (1 year) and week 104 (follow-up)
  Change from baseline (week 0) on World Health Organization Quality of Life Questionnaire - BREF (WHOQoL-BREF) scale at week 52 (1 year) and 104 (follow-up). Range 0-100. Higher score indicate better quality of life.
Change in Research and Development (RAND-36)/Short Form health survey (SF-36) (quality of life) | Week 0 (baseline), week 52 (1 year) and week 104 (follow-up)
  Change from baseline (week 0) on RAND-36/SF-36 scale at week 52 (1 year) and 104 (follow-up). Range 0-100. Higher score indicate better quality of life.
System Usability (SUS) | week 104 (follow-up)
  Usability of the Slow-SPEED-NL application assessed by the Dutch version of the System Usability Scale (SUS) at week 52 (year 1) and week 104 (follow-up). Range 0-100. Higher score indicate better usability.
Barriers and motivators to engage in physical activity | Week 0 (baseline) and week 104 (follow-up)
  Barriers and motivators to engage in physical activity reported on a self-developed questionnaire
Change in phenoconversion neurodegenerative disease | Week 0 (baseline) and week 104 (follow-up)
  Change from baseline (week 0) on phenoconversion in Parkinson's Disease (PD), Lewy body dementia (LBD) and multiple system atrophy (MSA). Higher scores indicate more phenoconversion.
Change in step count on a group level (compliance) | Week -4 until 0 (baseline) compared to week 0-26, week 26-52, week 52-78, week 78-104
  Change from week -4 until 0 (baseline period) mean step count per day compared to mean step count in 6 month periods. Mean step count per day will be calculated from 4-week periods. Scored as number of participants able to increase step count per day 0-25%, 26-50%, 51-75%, 76-100% relative to their own baseline measure
Change in moderate to vigorous physical activity per day on a group level (compliance) | Week -4 until 0 (baseline) compared to week 0-26, week 26-52, week 52-78, week 78-104
  Change from week -4 until 0 (baseline period) number of minutes exerting (minimally) ≥ 64% of maximum heart rate in 6 month periods. Mean minutes per day will be calculated from 4-week periods. Scored as number of participants to increase 0-25%, 26-50%, 51-75%, 76-100% relative to their own baseline measure
Number of completed step week goals on a group level (compliance) | Week 0 (baseline) and week 104 (follow-up)
  Total number of completed step count week goals
Number of completed aerobic activity (MVPA intensity) week goals on a group level (compliance) | Week 0 (baseline) and week 104 (follow-up)
  Total number of completed aerobic activity (MVPA intensity) week goals
Number of drop-outs on a group level (retention rate) | Week 0 (baseline), week 26, week 52, week 78, week 104 (follow-up)
  Number of drop-outs throughout the study
Number of interactions with Slow-SPEED app on a group level | Week 0 (baseline), week 26, week 52, week 78, week 104 (follow-up)
  Total times opening the app
Number of completed questionnaires on group level (completeness of digital assessments) | Week 0 (baseline), week 52, week 104 (follow-up)
  Number of completed questionnaires
Number of smartwatch data points on group level (completeness of digital assessments) | Week 0 (baseline), week 26, week 52, week 78, week 104 (follow-up)
  Number of data points received for each selected smartwatch parameter
Total smartwatch wear time on group level (completeness of digital assessments) | Week 0 (baseline), week 26, week 52, week 78, week 104 (follow-up)
  Total smartwatch wear time
Number of Roche PD Research mobile application data points on group level (completeness of digital assessments) | Week 0 (baseline), week 6, week 12, week 18, week 24, week 30, week 36, week 42, week 48, week 54, week 60, week 66, week 72, week 78, week 84, week 90, week 96, week 102
  Number of data points received

CONTACTS AND LOCATIONS:
Overall Officials: Sirwan KL Darweesh, PhD, Principal Investigator — Radboudumc Department of Neurology
Locations (1):
- Radboud University Medical Center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
We will make relevant anonymised data available in a database.
Supporting Information: Study Protocol
Time Frame: We will make relevant anonymised data available in a database after publication of the main results of our trial.
Access Criteria: Researchers who are interested in re-use of the data are asked to contact the central contact person for permission.